CLINICAL TRIAL: NCT00523094
Title: Vibration Response Imaging (VRI) in Patients That Are Candidates for Undergoing Pulmonary Operation Procedure
Status: Suspended | Type: Observational
Why Stopped: Enrollment was too slow and principal investigator moved to another country
Sponsor: Deep Breeze (Industry)
Responsible Party: Merav Gat/VP Clinical Affairs, Deep Breeze
Other Study IDs: DB032
Record Dates: First submitted 2007-08-29; First posted 2007-08-30 (Estimated); Last update posted 2009-06-16 (Estimated); Status verified 2009-06

CONDITIONS: Emphysema; Cancer
MeSH Terms: conditions — Emphysema; Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The primary objective of this study is to estimate the accuracy of the pre-operative VRI quantitative results versus the gold standard pre-operative perfusion scan.

The secondary objective is to assess the correlation of the predicted post-operative lung function with the observed post-operative lung function (forced expiratory volume in 1 second [FEV1] and diffusing capacity of the lung for carbon monoxide [DLCO]) in patients who underwent surgical resection.

DETAILED DESCRIPTION:
Pre lung operation candidates for procedures such as lung volume reduction surgery (LVRS), lung resection, bullectomy and lung transplant are frequently evaluated for differential lung function by a semi quantitative lung scintigraphy. VRI may offer the same differential lung function information for the physician without the risks, time and patient discomfort of lung scintigraphy in the treating physician office.

Moreover, VRI may provide a safe, quick and simple method to measure "split function" in lung cancer patients who are candidates for lung surgery. Thus eliminating the safety and complexity issue related with the current ventilation perfusion "split function" methods.

In addition the VRI may aid in achieving the goal of developing strategies to reduce risk and maximize the number of patients that can benefit from surgical therapy.

ELIGIBILITY:
Inclusion Criteria:

1. Able and willing to read, understand, and provide written informed consent;
2. Male or female in the age range of 18-80 years;
3. Patients who were referred to perform perfusion scan for pre lung surgery evaluation such as LVRS, thoracotomy, bullectomy and lobectomy.
4. Body mass index (BMI) > 21.

Exclusion Criteria:

1. Chest wall deformation;
2. Spine deformation (including scoliosis);
3. Hirsutism;
4. Potentially contagious skin lesion on the back;
5. Skin lesion that would interfere with sensor placement; (Keloids)
6. Cardiac pacemaker or implantable defibrillator;

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients evaluated for lung surgery who will undergo perfusion scan
Sampling Method: Non-Probability Sample
Enrollment: 75 (Estimated)
Dates: Start 2007-09; Study Completion 2008-07 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Atul C. Mehta, M.D, Principal Investigator — The Cleveland Clinic
Locations (1):
- Cleveland Clinic, Cleveland, Ohio, United States

REFERENCES:
- [Background] Benditt JO. Surgical therapies for chronic obstructive pulmonary disease. Respir Care. 2004 Jan;49(1):53-61; discussion 61-3. PMID 14733622
- [Background] Gurney JW. Pathophysiology of obstructive airways disease. Radiol Clin North Am. 1998 Jan;36(1):15-27. doi: 10.1016/s0033-8389(05)70005-1. PMID 9465866
- [Background] Salzman SH. Can CT measurement of emphysema severity aid patient selection for lung volume reduction surgery? Chest. 2000 Nov;118(5):1231-2. doi: 10.1378/chest.118.5.1231. No abstract available. PMID 11083665
- [Background] Corris PA, Ellis DA, Hawkins T, Gibson GJ. Use of radionuclide scanning in the preoperative estimation of pulmonary function after pneumonectomy. Thorax. 1987 Apr;42(4):285-91. doi: 10.1136/thx.42.4.285. PMID 3616987
- [Background] Arcasoy SM, Kotloff RM. Lung transplantation. N Engl J Med. 1999 Apr 8;340(14):1081-91. doi: 10.1056/NEJM199904083401406. No abstract available. PMID 10194239
- [Background] Hardoff R, Steinmetz AP, Krausz Y, Bar-Sever Z, Liani M, Kramer MR. The prognostic value of perfusion lung scintigraphy in patients who underwent single-lung transplantation for emphysema and pulmonary fibrosis. J Nucl Med. 2000 Nov;41(11):1771-6. PMID 11079482
- [Background] Cooper JD, Billingham M, Egan T, Hertz MI, Higenbottam T, Lynch J, Mauer J, Paradis I, Patterson GA, Smith C, et al. A working formulation for the standardization of nomenclature and for clinical staging of chronic dysfunction in lung allografts. International Society for Heart and Lung Transplantation. J Heart Lung Transplant. 1993 Sep-Oct;12(5):713-6. PMID 8241207
- [Background] Kristersson S, Lindell SE, Svanberg L. Prediction of pulmonary function loss due to pneumonectomy using 133 Xe-radiospirometry. Chest. 1972 Dec;62(6):694-8. doi: 10.1378/chest.62.6.694. No abstract available. PMID 4635418
- [Background] Olsen GN, Block AJ, Tobias JA. Prediction of postpneumonectomy pulmonary function using quantitative macroaggregate lung scanning. Chest. 1974 Jul;66(1):13-6. doi: 10.1378/chest.66.1.13. No abstract available. PMID 4846113
- [Background] Ali MK, Mountain CF, Ewer MS, Johnston D, Haynie TP. Predicting loss of pulmonary function after pulmonary resection for bronchogenic carcinoma. Chest. 1980 Mar;77(3):337-42. doi: 10.1378/chest.77.3.337. PMID 7357934
- [Background] Ali MK, Ewer MS, Atallah MR, Mountain CF, Dixon CL, Johnston DA, Haynie TP. Regional and overall pulmonary function changes in lung cancer. Correlations with tumor stage, extent of pulmonary resection, and patient survival. J Thorac Cardiovasc Surg. 1983 Jul;86(1):1-8. PMID 6865454
- [Background] Kearney DJ, Lee TH, Reilly JJ, DeCamp MM, Sugarbaker DJ. Assessment of operative risk in patients undergoing lung resection. Importance of predicted pulmonary function. Chest. 1994 Mar;105(3):753-9. doi: 10.1378/chest.105.3.753. PMID 8131537
- [Background] Markos J, Mullan BP, Hillman DR, Musk AW, Antico VF, Lovegrove FT, Carter MJ, Finucane KE. Preoperative assessment as a predictor of mortality and morbidity after lung resection. Am Rev Respir Dis. 1989 Apr;139(4):902-10. doi: 10.1164/ajrccm/139.4.902. PMID 2930068